CLINICAL TRIAL: NCT07022990
Title: Promoting Healthy Aging Among WTC Responders: Frailty Trajectories And Intervention Strategies
Brief Title: Improving Medication Management in World Trade Center Responders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Fred Ko, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY-22-00737; 21-2114-00001 (Other Grant/Funding Number: National Institute for Occupational Safety and Health); U01OH012473 (NIH)
Record Dates: First submitted 2025-06-08; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Polypharmacy
Keywords: Deprescribe; Medication management
MeSH Terms: interventions — Deprescriptions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- World Trade Center (WTC) Responders (Experimental): World Trade Center (WTC) rescue and recovery workers (responders).
  Interventions: Other: Educational brochure for deprescribing

INTERVENTIONS:
Other: Educational brochure for deprescribing — Study participant will be provided information (i.e., educational brochure) about one of the five medication classes participants may be taking that are known to have potential side effects for older adults: proton pump inhibitors (PPIs), benzodiazepine (BZs) and non-benzodiazepine sedative hypnotics ("Z-drugs"), first-generation antihistamines (FGA), and skeletal muscle relaxants (SMR) to determine their necessity.

SUMMARY:
By 2030, the majority of World Trade Center (WTC) rescue and recovery workers (responders) will be aged 65 and over and at risk for aging-related conditions and consequences including the concurrent use of five or more medications (i.e., polypharmacy). The purpose of this research study is to investigate an educational approach targeting polypharmacy through de-prescribing unnecessary and burdensome medications via the support of informed discussions between WTC responders and their prescribing physicians.

DETAILED DESCRIPTION:
De-prescribing is the act of reducing or stopping medications that are no longer necessary or may cause harm, to reduce adverse drug reactions and ensure the safety of patients. Polypharmacy is the simultaneous use of five or more medications. Through education brochures and discussions about potential side effects of medications, the research team will see whether these approaches lead to discussions between a study participant (WTC responder) and the prescribing physician, to make informed decisions about management of medications. Specifically, the participant will be provided information about one of the five medication classes they may be taking that are known to have potential side effects for older adults: proton pump inhibitors (PPIs), benzodiazepine (BZs) and non-benzodiazepine sedative hypnotics ("Z-drugs"), first-generation antihistamines (FGA), and skeletal muscle relaxants (SMR) to determine their necessity. To be clear, changes to medications will only be done under the guidance of the prescriber.

Study participants will be asked to complete baseline surveys that ask about beliefs and attitudes regarding medications and de-prescribing; review patient education brochure about a medication the participant is taking; discuss deprescribing options with the participant's prescriber; and complete a survey regarding acceptance of the deprescribing intervention and how this process may have affected the physician-patient relationship.

ELIGIBILITY:
Inclusion Criteria:

* A WTC responder already enrolled in the "Promoting Healthy Aging Among WTC Responders: Frailty Trajectories and Intervention Strategies" study cohort
* aged 50 years or older, and
* taking one of the five medication classes:

  * proton pump inhibitors (PPIs),
  * benzodiazepine (BZs) and
  * non-benzodiazepine sedative hypnotics ("Z-drugs"),
  * first-generation antihistamines (FGA), and
  * skeletal muscle relaxants (SMR).

Exclusion Criteria:

* None

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-08 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Brief Medication Questionnaire 2 (BMQ2) | 6 months after study enrollment
  Brief Medication Questionnaire 2 (BMQ2) to measure participants feel/views about Z Drugs, Skeletal Muscle Relaxants, Proton Pump Inhibitors and Benzodiazepines. Min scale: Strongly Agree - Max scale: Strongly Disagree. Higher score means patient strongly disagrees with the extent medications makes them feel/views about their medication.

SECONDARY OUTCOMES:
Patient-reported Attitudes Towards Deprescribing (rPATD) | 6 months after study enrollment
  The Revised Patients' Attitudes Towards Deprescribing (rPATD) questionnaire consists of 22 items divided into five subscales: perceived burden of medication taking, concerns about stopping the medication, belief in appropriateness of medication use (harms/benefits), level of involvement/knowledge of medications, and global questions. Each item is rated on a 5-point Likert scale: 5 = strongly agree, 4 = agree, 3 = unsure, 2 = disagree, and 1 = strongly disagree. The total score ranges from 22 to 110, with higher scores indicating greater perceived burden, concern, involvement, or agreement with global questions. Subscale scores are: perceived burden (5 items, 5-25), concerns about stopping (5 items, 5-25), belief in appropriateness (5 items, 5-25, reversed), involvement/knowledge (5 items, 5-25), and global questions (2 items, 2-10). Higher scores indicate greater concern or involvement, with reversed scoring for the belief in appropriateness subscale.

CONTACTS AND LOCATIONS:
Overall Officials: Fred Ko, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal. To achieve aims in the approved proposal. Specify Other Mechanism Data will be provided directly to researchers who have approval under the direction of WTC General Responder Data Center and study PIs.